CLINICAL TRIAL: NCT04128943
Title: Electronic Patient-reported Outcome Monitoring in Patients With Aplastic Anemia and Paroxysmal Nocturnal Hemoglobinuria - a Pilot Study
Brief Title: Electronic Patient-reported Outcome Monitoring in Aplastic Anemia and Paroxysmal Nocturnal Hemoglobinuria
Acronym: ePRO-AA-PNH
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ProPatient foundation of the University Hospital Basel (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-01563; me18Drexler
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Aplastic Anemia; Paroxysmal Nocturnal Hemoglobinuria
Keywords: electronic patient-reported outcomes; electronic health (eHealth) technology; app utilization; ePRO application
MeSH Terms: conditions — Anemia, Aplastic; Hemoglobinuria, Paroxysmal | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: symptom questionnaire — A weekly filled in symptom questionnaire for reported symptoms of AA and/or PNH (yes/no, grade, date). Grading according to current grading systems (Common Terminology Criteria for Adverse Events,CTCAE).
  Data collection and processing via the ePRO application by Kaiku Health Ltd
Other: recording of vital signs — Record function for vital parameters (blood pressure, temperature and pulse); Data collection and processing via the ePRO application by Kaiku Health Ltd
Other: European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 questionnaire — The EORTC QLQ-C30 incorporates nine multi-item scales: five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties). All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Other: interview — Interview with the patients and responsible medical team by phone or during hospital visit about functional problems regarding the application (duration: 15-30 min) to avoid incorrect use of the application, at week 3 and month 3 and month 6

SUMMARY:
Aplastic anemia (AA) and paroxysmal nocturnal hemoglobinuria (PNH) are interrelated and very rare diseases. Therefore, little data about clinical characteristics, especially the variety of symptoms in the course of the respective disease are available. As a consequence, patients may be left on their own between infrequent follow-ups at a specialist center. A web-based symptom-monitoring application can support selfmanagement and patient empowerment and promotes a patient- centered interdisciplinary team approach in the context of a "disease management program". This pilot study is to investigate usability and feasibility of the electronic Patient-Reported Outcome (ePRO) application in AA/PNH by assessing recruitment, app utilization, data collection, functionality, acceptability after using and working with the ePRO application.

ELIGIBILITY:
Inclusion Criteria:

* AA (acquired and hereditary) and/or PNH patients
* Minimal level of computer literacy with prior email experience and access to an Internet connection

Exclusion Criteria:

* Mental alteration or psychiatric disease that can compromise written informed consent or adherence to the protocol and monitoring of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated at the University Hospital Basel for AA and/or PNH
Sampling Method: Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
recruitment with the ePRO application (number) | Day 1= Day of inclusion
  Analyses of usability of the ePRO application by assessing recruitment with the ePRO application
usability of the ePRO application | Weekly assessments from Day 1= Day of inclusion until Day 180 (+/- 7 days) = last day of testing phase
  Descriptive analyses of usability of the ePRO application by assessing data collection with the ePRO application
acceptability of the ePRO application | Weekly assessments from Day 1= Day of inclusion until Day 180 (+/- 7 days) = last day of testing phase
  Descriptive analyses of acceptability of the ePRO application by assessing app utilization

SECONDARY OUTCOMES:
Change in quality of life assessed by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C30 questionnaire (EORTC QLQ-C30 questionnaire) | at day 1= Day of inclusion and at day 180 (+/- 7 days) = last day of testing phase
  Change in quality of life assessed by the EORTC QLQ-C30 questionnaire. The EORTC QLQ-C30 incorporates nine multi-item scales: five functional scales (Physical, Role, Cognitive, Emotional and Social Functioning); three symptom scales (Fatigue, Pain and Nausea/Vomiting); and a Global Health Status/QoL scale. Six single item scales are also included (Dyspnoea, Insomnia, Appetite Loss, Constipation, Diarrhoea and Financial Difficulties). All of the scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Drexler, Dr. med, Principal Investigator — Division of Hematology, University Hospital Basel
Locations (1):
- Division of Hematology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Banziger S, Weisshaar K, Arokoski R, Gerull S, Halter J, Rovo A, Bargetzi M, Goede JS, Senft Y, Valenta S, Passweg JR, Drexler B. Feasibility of electronic patient-reported outcome monitoring and self-management program in aplastic anemia and paroxysmal nocturnal hemoglobinuria-a pilot study (ePRO-AA-PNH). Ann Hematol. 2023 Jan;102(1):199-208. doi: 10.1007/s00277-022-05012-5. Epub 2022 Nov 3. PMID 36326854